CLINICAL TRIAL: NCT04753515
Title: Comparison Between Dexmedetomidine and Propofol for Sedation When Combined With Midazolam and Remifentanil During Awake Endotracheal Intubation: A Randomized Double-blind Controlled Study
Brief Title: Dexmedetomidine Versus Propofol for Sedation During Awake Endotracheal Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, SanQing Jin, professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2020154
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Sedation; Intubation
Keywords: Awake tracheal Intubation
MeSH Terms: interventions — Midazolam; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group DMR (Active Comparator): dexmedetomidine combined with midazolam and remifentanil.
  Interventions: Drug: dexmedetomidine combined with midazolam and remifentanil.
- Group PMR (Active Comparator): propofol combined with midazolam and remifentanil.
  Interventions: Drug: propofol combined with midazolam and remifentanil.

INTERVENTIONS:
Drug: dexmedetomidine combined with midazolam and remifentanil. — Patients in this group will receive a bolus of midazolam 0.03 mg/kg intravenously, and then a loading dose of 0.5 mcg/kg remifentanil and 0.5 mcg/kg dexmedetomidine over 5 min via separate syringe pumps.
  Other Names: dexmedetomidine-midazolam-remifentanil
  Arms: Group DMR
Drug: propofol combined with midazolam and remifentanil. — Patients in this group will receive a bolus of midazolam 0.03 mg/kg intravenously, and then a loading dose of 0.5 mcg/kg remifentanil and 0.33 mg/kg propoful over 5 min via separate syringe pumps.
  Other Names: propofol-midazolam-remifentanil
  Arms: Group PMR

SUMMARY:
The purpose of this study is to compare the sedation effect of dexmedetomidine and propofol when they are both combined with midazolam and remifentanil during awake endotracheal intubation.

DETAILED DESCRIPTION:
Awake intubation is one of the best strategy guaranteed by the American Society of Anesthesiologists (ASA) guidelines for the management of patients with anticipated difficult airways. Hemodynamic stability, optimal intubating conditions, patients' comfort, amnesia and preservation of patents' spontaneous respiration are critical for awake intubation. Sedation is one of the key elements for this technique. Intravenous midazolam, propofol, dexmedetomidine and remifentanil are commonly used as sedatives during awake intubation. These agents are not preferred to be used alone but in combination with each other for the purpose of minimizing their respective side effects. The aim of this randomized controlled trial is to compare the safety and effectiveness of dexmedetomidine versus propofol for sedation during awake endotracheal intubation when they are both combined with midazolam and remifentanil.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 Years old;
2. scheduled for elective surgery under general anesthesia with oral tracheal intubation;
3. The American Society of Anesthesiologists(ASA) grade is I or II, and the cardiac function is 1-2;
4. Body mass index (BMI) 18-30 kg/m2.

Exclusion Criteria:

1. Patients have severe cardiac diseases (cardiac function grading greater than grade 3/arrhythmia including sick sinus syndrome, atrial fibrillation, atrial flutter, atrioventricular block, frequent ventricular premature, multiple ventricular premature, ventricular premature R on T, ventricular fibrillation and ventricular flutter/acute coronary syndrome) or respiratory failure or hepatic failure or renal failure;
2. body mass index (BMI) ≥30 kg/m2 or <18 kg/m2;
3. Patients with poor blood pressure control (receive regular antihypertensive medical treatment but still have systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 90 mmHg);
4. Patients with a higher risk of reflux and aspiration, such as full stomach, gastrointestinal obstruction, gastroparesis, and pregnant women;
5. Patients have schizophrenia, epilepsy, Parkinson's disease, intellectual disability, hearing impairment.;
6. Patients who take sedative and analgesic drugs for a long time;
7. Patients who are allergic to propofol, dexmedetomidine, midazolam or remifentanil
8. Patients who are expected to be difficult to intubate;
9. Patients who are participating in other clinical trials, or who refuse to sign informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
blood pressure | During the procedure of general anesthesia induction, expected an average of 20 min
  systolic blood pressure (SBP), diastolic blood pressure (DBP), and mean blood pressure (MBP) shown in the monitor.

SECONDARY OUTCOMES:
intubation condition score | During the procedure of general anesthesia induction, expected an average of 20 min
  Assessment of the intubation condition according to the scale of the modified Erhan's intubation condition score which includes jaw relaxation, laryngoscopy, vocal cord position, and patient's response (coughing, limb movement) to intubation and inflation of the intubation tube cuff.

OTHER OUTCOMES:
degree of coughing | During the procedure of general anesthesia induction, expected an average of 20 min.
  Grade assessment of coughing during the peri-intubation period (1 = No cough and limb activity, 2 = Intermittent cough with slight activity of chest and abdomen, 3 = Continuous cough with large amplitude activity of chest and abdomen, no limb activity, 4 = Continuous cough with large amplitude activity of chest and abdomen and limbs)
heart rate | During the procedure of general anesthesia induction, expected an average of 20 min.
  Heart rate shown in the monitor
pulse oxygen saturation (SpO2) | During the procedure of general anesthesia induction, expected an average of 20 min.
  SpO2 shown in the monitor
level of recall | postoperative follow-up visit 24 hours after the operation, expected an average of 5 min.
  At the 24-h postoperative follow-up visit, patients will be interviewed to assess their recall of pre-anesthesia events, administration of topical anesthesia, endoscopy and intubation.
satisfaction score | postoperative follow-up visit 24 hours after the operation, expected an average of 5 min.
  At the 24-h postoperative follow-up visit, patients will be interviewed to assess their satisfaction about the procedure of awake intubation (1 = excellent, 2 = good, 3 = fair, 4 = poor).
adverse events | postoperative follow-up visit 24 hours after the operation, expected an average of 5 min.
  At the 24-h postoperative follow-up visit, patients will be interviewed to assess the adverse events related to endotracheal intubation (postoperative hoarseness or sore throat)

CONTACTS AND LOCATIONS:
Overall Officials: SanQing Jin, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apfelbaum JL, Hagberg CA, Caplan RA, Blitt CD, Connis RT, Nickinovich DG, Hagberg CA, Caplan RA, Benumof JL, Berry FA, Blitt CD, Bode RH, Cheney FW, Connis RT, Guidry OF, Nickinovich DG, Ovassapian A; American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Practice guidelines for management of the difficult airway: an updated report by the American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Anesthesiology. 2013 Feb;118(2):251-70. doi: 10.1097/ALN.0b013e31827773b2. No abstract available. PMID 23364566
- [Background] Zhou LJ, Fang XZ, Gao J, Zhangm Y, Tao LJ. Safety and Efficacy of Dexmedetomidine as a Sedative Agent for Performing Awake Intubation: A Meta-analysis. Am J Ther. 2016 Nov/Dec;23(6):e1788-e1800. doi: 10.1097/MJT.0000000000000319. PMID 26196522
- [Background] Cattano D, Lam NC, Ferrario L, Seitan C, Vahdat K, Wilcox DW, Hagberg CA. Dexmedetomidine versus Remifentanil for Sedation during Awake Fiberoptic Intubation. Anesthesiol Res Pract. 2012;2012:753107. doi: 10.1155/2012/753107. Epub 2012 Jul 16. PMID 22844277
- [Background] Xu T, Li M, Ni C, Guo XY. Dexmedetomidine versus remifentanil for sedation during awake intubation using a Shikani optical stylet: a randomized, double-blinded, controlled trial. BMC Anesthesiol. 2016 Aug 2;16(1):52. doi: 10.1186/s12871-016-0219-9. PMID 27484783
- [Background] Johnston KD, Rai MR. Conscious sedation for awake fibreoptic intubation: a review of the literature. Can J Anaesth. 2013 Jun;60(6):584-99. doi: 10.1007/s12630-013-9915-9. Epub 2013 Mar 20. PMID 23512191
- [Background] Park S, Choi SL, Nahm FS, Ryu JH, Do SH. Dexmedetomidine-remifentanil vs propofol-remifentanil for monitored anesthesia care during hysteroscopy: Randomized, single-blind, controlled trial. Medicine (Baltimore). 2020 Oct 23;99(43):e22712. doi: 10.1097/MD.0000000000022712. PMID 33120766